STUDY TITLE: DMID 11-0069

# Statistical Analysis Plan

| TRIAL FULL TITLE | A PHASE II RANDOMIZED AND CONTROLLED |
|---|---|
| | INVESTIGATION OF SIX WEEKS OF ORAL |
| | VALCANCICLOVIR THERAPY IN INFANTS AND CHILDREN |
| | WITH CONGENITAL CYTOMEGALOVIRUS INFECTION AND |
| | HEARING LOSS |
| | DMID Protocol Number: 11–0069 |
| EUDRACT NUMBER | |
| SAP VERSION | 2.0 |
| ISRCTN NUMBER | |
| SAP VERSION DATE | 14 August 2020 |
| TRIAL STATISTICIANS | Inmaculada Aban, PhD, Charity Morgan, PhD, Kalyani |
| | Peri, MS |
| TRIAL CHIEF | David Kimberlin, MD |
| INVESTIGATOR | |
| SAP AUTHOR | Inmaculada Aban, PhD; Charity Morgan, PhD, Kalyani |
| | Peri, MS, Jill Griffin |

# **Table of Contents**

| T | able | of Co | ontents | 2 |
|---|---|---|---|---|
| 1 | Α | bbrev | viations and Definitions | 4 |
| 2 | In | ntrodi | uction | 6 |
| | 2.1 | Pre | eface | 6 |
| | 2.2 | Pu | rpose of the analyses | 6 |
| 3 | St | tudy ( | Objectives and Endpoints | 6 |
| | 3.1 | Stı | udy Objectives | 6 |
| | 3.2 | En | dpoints | 6 |
| | 3.3 | De | rived variables | 8 |
| 4 | St | tudy l | Methods | 9 |
| | 4.1 | Ge | neral Study Design and Plan | 9 |
| | 4.2 | Eq | uivalence or Non-Inferiority Studies | .12 |
| | 4.3 | Ind | clusion-Exclusion Criteria and General Study Population | .13 |
| | 4.4 | Ra | ndomization and Blinding | 14 |
| | 4.5 | Stı | udy Variables | 15 |
| 5 | Sa | ample | e Size | 19 |
| 6 | G | enera | ıl Considerations | 19 |
| | 6.1 | Tir | ming of Analyses | 19 |
| | 6.2 | An | alysis Populations | 19 |
| | 6.3 | Co | variates and Subgroups | 20 |
| | 6.4 | Mi | ssing Data | 20 |
| | 6.5 | Int | erim Analyses and Data Monitoring | 20 |
| | 6 | .5.1 | Safety Review | 21 |
| | 6 | .5.2 | Stopping Rules | 21 |
| | 6 | .5.3 | Adjustment of Confidence Intervals and p-values | .22 |
| | 6 | .5.4 | Practical Measures to Minimize Bias | 23 |
| | 6 | .5.5 | Documentation of Interim Analyses | 23 |

| | 6.6 | Multi-center Studies | 23 |
|---|---|---|---|
| | 6.7 | Multiple Testing | 23 |
| 7 | Sı | ummary of Study Data | 23 |
| | 7.1 | Subject Disposition | 24 |
| | 7.2 | Protocol Deviations | 27 |
| | 7.3 | Demographic and Baseline Variables | 27 |
| | 7.4 | Degree of CMV Disease Involvement at Birth | 27 |
| | 7.5 | Concurrent Illnesses and Medical Conditions | 28 |
| | 7.6 | Prior and Concurrent Medications | 28 |
| | 7.7 | Treatment Compliance | 28 |
| 8 | Ef | ficacy Analyses | 29 |
| | 8.1 | Primary Efficacy Analysis | 29 |
| | 8.2 | Secondary Efficacy Analyses | 30 |
| 9 | Sa | afety Analyses | 31 |
| | 9.1 | Extent of Exposure | 32 |
| | 9.2 | Adverse Events | 32 |
| | 9.3 | Deaths, Serious Adverse Events and other Significant Adverse Events | 32 |
| | 9.4 | Pregnancies | 32 |
| | 9.5 | Clinical Laboratory Evaluations | 32 |
| | 9.6 | Other Safety Measures | 33 |
| 1 | 0 | Pharmacokinetics | 33 |
| 1 | 1 | Virology | 34 |
| 1 | 2 | Figures | 35 |
| 1 | 3 | Reporting Conventions | 35 |
| 1 | 4 | Technical Details | 36 |
| 1 | 5 | Summary of Changes to the Protocol | 37 |
| 1 | 6 | References | 37 |
| 1 | 7 | Listing of Tables and Listings Figures | 39 |

## 1 Abbreviations and Definitions

AE Adverse Event/Adverse Experience

AIC Akaike Information Criteria
ANC Absolute Neutrophil Count

AUC Area Under the Curve

BSER Brainstem Evoked Response

CASG Collaborative Antiviral Study Group

CL/F Oral Clearance CMV Cytomegalovirus

CNS Central Nervous System
Cobs Observed Concentration
Cpred Predicted Concentration

CRF Case Report Form

CROMS Clinical Research Operations and Management Support

CSF Cerebrospinal Fluid

CU Central Unit

DAIDS The United States Division of AIDS

DCC Data Coordinating Center

DMID Division of Microbiology and Infectious Diseases, NIAID, NIH, DHHS

DSMB Data and Safety Monitoring Board

eDES Electronic Data Entry System

FDA Food and Drug Administration, USA

GCV Ganciclovir

GEE Generalized Estimating Equations
HEENT Head, ears, eyes, nose and throat
HIV Human Immunodeficiency Virus

IA Independent Audiologist

IPAM Integrated Pharmacokinetic Adherence Measure

ITT Intent to Treat
IV Intravenous
Ka Absorption Rate

Ke Elimination Constant

kg Kilogram L Liter

L/hr Liter Per Hour
L Log Likelihood

MedDRA Medical Dictionary for Regulatory Activities

STUDY TITLE: DMID 11-0069

#### Statistical Analysis Plan

mg Milligram

MLEM Maximum Likelihood Estimation Maximization

N Number (typically refers to subjects)

N/A Not applicable

NIAID National Institute of Allergy and Infectious Diseases, NIH, DHHS

STUDY TITLE: DMID 11-0069

NIH National Institutes of Health

OAE Otoacoustic Emissions

PCR Polymerase Chain Reaction

PK Pharmacokinetic
PP Per-protocol

SAE Serious Adverse Event//Serious Adverse Experience

SAP Statistical Analysis Plan

Scr Serum creatinine
SE Standard error

SNHL Sensorineural Hearing Loss

 $T_{1/2}$  Time of Half life

UAB University of Alabama at Birmingham

V/F Volume of Distribution

VGCV Valganciclovir

VRA Visual Reinforcement Audiometry

WBC White Blood Cell

## 2 Introduction

#### 2.1 Preface

This study is a Phase II, international, multi-center, double-blind, placebo-controlled evaluation of six weeks of valganciclovir treatment for children (up to 4 years of age) with virologically-confirmed congenital CMV infection and hearing loss. In order for the treatment arms of the trial to remain blinded, a valganciclovir placebo will be utilized, as described below. Patients meeting inclusion/exclusion criteria will be offered enrollment onto the trial.

STUDY TITLE: DMID 11-0069

# 2.2 Purpose of the analyses

These analyses will evaluate whether six weeks of antiviral therapy can stabilize hearing deterioration in older infants, toddlers, and young children who have developed CMV-associated hearing loss.

# 3 Study Objectives and Endpoints

# 3.1 Study Objectives

(ICH E3; 8.)

- To assess whether a six week course of oral valganciclovir can stabilize the hearing of children with congenital CMV infection who present with hearing loss.
- To measure CMV viral load in blood, urine, and saliva as a function of systemic exposure to ganciclovir (active metabolite of valganciclovir).
- To define the safety and tolerability of valganciclovir in enrolled subjects.
- To define the pharmacokinetics of ganciclovir (metabolite) following administration valganciclovir (prodrug) in enrolled subjects.

# 3.2 Endpoints

(ICH E9; 2.2.2)

**Primary Endpoint** 

Change in total ear hearing assessments (improved + no change versus other) between Baseline and Study Month 6

#### **Secondary Endpoints**

- 1. Change in best ear hearing assessments [improved + no change (normal to normal) versus other; improved versus other; worse + no change (abnormal to abnormal) versus other; and worse versus other] between Baseline and Study Month 6
- 2. Change in total ear hearing assessments (improved versus other; worse + no change (abnormal to abnormal) versus other; and worse versus other) between Baseline and Study Month 6
- 3. Detection of viruria by PCR six weeks and six months after trial entry
- 4. The quantitative log reduction in viruria detected after 6 weeks of therapy
- 5. Detection of viremia by PCR six weeks and six months after trial entry
- 6. The quantitative log reduction in viremia detected after 6 weeks of therapy
- 7. Detection of CMV in saliva by PCR six weeks and six months after trial entry
- 8. The quantitative log reduction in CMV viral load in saliva detected after 6 weeks of therapy
- 9. Correlation of change in viral load with change in total ear and best ear hearing at 6 months
- 10. Incidence of unanticipated medically attended visits occurring from Study Day 1 through two weeks following the last dose of study drug
- 11. Incidence of adverse events which lead to permanent discontinuation of valganciclovir therapy or have an unresolved outcome

#### **Tertiary Endpoints**

1. Blood concentrations of ganciclovir after administration of valganciclovir

#### 3.3 Derived variables

The primary efficacy assessment will be change in total ear hearing assessment between baseline and 6 months post enrollment. Categories used for hearing assessment of each ear for each time point will be normal hearing, mild hearing loss, moderate hearing loss, and severe hearing loss. Baseline and 6 month hearing categories will be compared and the change in each ear will be categorized into binary outcomes: Improved or no change versus Other (i.e., worsened) Note that the total ear assessment at each time point will be provided by the Independent Audiologist and entered in the database following the rules below and the information provided by the audiology reports.

STUDY TITLE: DMID 11-0069

In the model-based analyses, the "no change" category will be broken down into "Protected: normal to normal" as one category and "No Change: same degree of hearing loss at Baseline and Study Month 6" as another category. The rationale behind this is that if one is interested in the improvement of hearing loss, a subject that has normal hearing at baseline cannot improve further. Hence from an efficacy analysis point of view, the "Protected: normal to normal" can be viewed as protective effect of the drug from hearing deterioration. This analysis approach will be similar to the analysis of the previous CASG study that established the efficacy of 6 weeks of IV GCV in symptomatic congenital CMV disease with CNS involvement.

Analysis of actual viral load will be done using log base 10 transformation. Undetectable viral load value will be replaced by a value of 10. A summary measure of the viral load over time—will be calculated two ways. The first approach considers all time points available by calculating the average area under the curve (AUC) (trapezoidal rule) applied to the log base 10 viral load. Average is based on the maximum period of time with viral load data for a given subject. To illustrate, if the calculated AUC for log10 VL for a given subject is 200 from baseline to Day 70, then average AUC is 200/70=2.86. Taking average AUC will enable us to use and compare data from subjects who did not have viral load values at the later time due to dropping out early, for example, with subjects with complete viral load data. The second approach is to take using difference between Month 6 and baseline log10 VL. The last visit with available VL will be used for those without Month 6 VL. Section 11 contains more details on Viral Load analyses.

PK data analyses and computations of PK-related derived variables are detailed in Section 10.

# 4 Study Methods

# 4.1 General Study Design and Plan

(ICH E3;9)

The current study evaluates whether six weeks of antiviral therapy can stabilize hearing deterioration in older infants, toddlers, and young children who have developed CMV-associated hearing loss. This study is a Phase II, international, multi-center, double-blind, placebo-controlled evaluation of six weeks of valganciclovir treatment for children (up to 4 years of age) with virologically-confirmed congenital CMV infection and hearing loss.

STUDY TITLE: DMID 11-0069

Patients meeting inclusion/exclusion criteria will be offered enrollment into the trial. Randomization on the study occurs when the diagnosis of congenital CMV infection is confirmed, and the subject is then assigned to receive either 6 weeks of oral valganciclovir or 6 weeks of placebo. Study subjects will be stratified according to age at randomization (1 through 11 months, 12 through 23 months, 24 through 35 months, and  $\geq$  36 months) and CMV involvements (symptomatic and asymptomatic at birth) as a marker of disease severity. An independent Data and Safety Monitoring Board (DSMB) will oversee the conduct of the trial. During the course of their oversight, they may request to have access to unblinded data.

The target sample size is 54 subjects (27 in each arm). Up to 20% over-enrollment will be allowed to replace subjects who drop-out or who have inadequate audiology assessments. The primary endpoint will be change in total ear hearing assessments (improved + no change versus other) between baseline and 6 months. Secondary and tertiary endpoints will be assessments of other measures of hearing outcomes; detection of viruria, viremia, and CMV in saliva by PCR six weeks and six months after trial entry; the quantitative log reduction in viruria, viremia, and CMV viral load in saliva detected after six weeks of therapy; correlation of change in viral load with change in total ear and best ear hearing at six months; incidences of unanticipated medically attended visits and adverse events which lead to permanent discontinuation of valganciclovir therapy or have an unresolved outcome; and assessments of blood concentration of ganciclovir after administration of valganciclovir. Stopping rules will be employed in order to limit exposure of study subjects to a potentially unacceptable treatment.

Figure 1: Schematic of Study Design



Timing of study visits (days, months) for collection of urine, saliva, and blood (together with safety laboratory measurements at Study Days 1, 14, 28, 42 and 70)

During the 6 week treatment period and for 4 week thereafter, study subjects will be followed every two weeks for 6 weeks. Subjects will then be seen a month after the end of the treatment period, then at 4 and 6 months after randomization. During the 6 week treatment period and at the 1 month post treatment period, safety labs will be checked and adverse events will be assessed. The dose of study medication will be adjusted for weight change at each of these study treatment visits, hence collection of growth parameters at each of the treatment visits. Whole blood will be obtained for CMV viral load at each of these visits as well. Hearing outcomes will be assessed at baseline and 6 months. Changes in whole blood viral load measurements will be correlated with hearing outcome.

## Safety Reviews and Halting Rules

Halting rules for this study therefore have been constructed to interrupt study enrollment if an excessive number of subjects are experiencing neutropenia. Assuming that 75% of subjects receiving ganciclovir developed Grade 3 or 4 neutropenia and given that randomization is expected to be balanced between those in study drug and those in placebo, the stopping rule will be based on assuming that the overall event rate for all study participants (i.e., placebo and active subjects combined) is 37.5%. Therefore, study enrollment will be stopped and an ad hoc review will be performed if a significantly higher proportion (37.5%) of subjects in this study experience Grade 3 or Grade 4 neutropenia, as detailed in the following table:

X of the first Y subjects enrolled have Grade 3 or Grade 4 neutropenia, according to the table below. The stopping rules are based on the upper tail probabilities of the cumulative binomial with probability of an event set at 0.375. The cut-off numbers were determined by obtaining the largest value such that the tail probability is less than but closest to 0.05.

| Number<br>enrolled (Y) | Stop/Investigate<br>when number with<br>events equals this<br>number (X) | Probability of<br>observing X or<br>more events<br>assuming<br>p=0.375 | Number<br>enrolled (Y) | Stop/Investigate when<br>number with events<br>equals this number (X) | Probability of<br>observing X or<br>more events<br>assuming<br>p=0.375 |
|---|---|---|---|---|---|
| 4 | 4 | 0.020 | 30 | 17 | 0.025 |
| 5 | 5 | 0.007 | 31 | 17 | 0.037 |

| 6 | 5 | 0.031 | 32 | 18 | 0.024 |
|----|----|-------|----|----|-------|
| 7 | 6 | 0.013 | 33 | 18 | 0.034 |
| 8 | 6 | 0.036 | 34 | 18 | 0.048 |
| 9 | 7 | 0.017 | 35 | 19 | 0.032 |
| 10 | 7 | 0.038 | 36 | 19 | 0.044 |
| 11 | 8 | 0.019 | 37 | 20 | 0.030 |
| 12 | 8 | 0.039 | 38 | 20 | 0.041 |
| 13 | 9 | 0.021 | 39 | 21 | 0.028 |
| 14 | 9 | 0.039 | 40 | 21 | 0.038 |
| 15 | 10 | 0.021 | 41 | 22 | 0.026 |
| 16 | 10 | 0.037 | 42 | 22 | 0.035 |
| 17 | 11 | 0.021 | 43 | 22 | 0.047 |
| 18 | 11 | 0.036 | 44 | 23 | 0.032 |
| 19 | 12 | 0.021 | 45 | 23 | 0.043 |
| 20 | 12 | 0.034 | 46 | 24 | 0.030 |
| 21 | 13 | 0.020 | 47 | 24 | 0.040 |
| 22 | 13 | 0.033 | 48 | 25 | 0.028 |
| 23 | 13 | 0.050 | 49 | 25 | 0.037 |
| 24 | 14 | 0.031 | 50 | 25 | 0.048 |
| 25 | 14 | 0.046 | 51 | 26 | 0.034 |
| 26 | 15 | 0.029 | 52 | 26 | 0.044 |
| 27 | 15 | 0.043 | 53 | 27 | 0.032 |
| 28 | 16 | 0.027 | 54 | 27 | 0.041 |
| 29 | 16 | 0.040 | | | |

In addition to the continual assessment of serious adverse events leading to permanent discontinuation from protocol, the DSMB may request for unblinded safety profile listings.

# 4.2 Equivalence or Non-Inferiority Studies

(ICH E3; 9.2, 9.7.1, 11.4.2.7. ICH E9; 3.3.2)

Not applicable

# **4.3 Inclusion–Exclusion Criteria and General Study Population** (ICH E3;9.3. ICH E9;2.2.1)

Male and female infants from 1 month through 3 years of age (up to 4th birthday) with sensorineural hearing loss will be eligible for enrollment. Following confirmation of inclusion/exclusion criteria and the signing of informed consent, the subject's Guthrie card will be retrieved and tested for CMV DNA by PCR unless there is a virologically confirmed diagnosis of congenital CMV infection made within the first 30 days of life. Inclusion criteria were selected to ensure the inclusion of those subjects with congenital CMV disease. Exclusion criteria were selected to limit confounders for safety and efficacy. Renal insufficiency was an exclusion criterion because the active moiety, GCV, is renally cleared and a neonate's renal system is not fully developed. The study population is consistent with those patients seen in clinical practice and who receive IV GCV as standard of care to treat symptomatic congenital CMV.

#### **Inclusion Criteria**

- Signed informed consent from parent(s) or legal guardian(s)
- Sensorineural hearing loss (≥ 21dB in one or both ears, documented within 12 weeks prior to study entry)
- Children from 1 month through 3 years of age (up to the 4th birthday)

#### **Exclusion Criteria**

- Imminent demise
- Profound sensorineural hearing loss (> 90dB) in both ears
- Patients receiving other antiviral agents or immune globulin
- Gastrointestinal abnormality which might preclude absorption of an oral medication (e.g., a history of necrotizing enterocolitis)
- Documented renal insufficiency, as noted by a creatinine clearance < 10 mL/min/1.73m<sup>2</sup> at time of study enrollment
- Breastfeeding from mother who is receiving ganciclovir, valganciclovir, foscarnet, cidofovir, or maribavir
- Infants known to be born to women who are HIV positive (but HIV testing is not required for study entry).
- Current receipt of other investigational drugs
- Previous receipt of ganciclovir or valganciclovir

- STUDY TITLE: DMID 11-0069
- Known hypersensitivity to ganciclovir, valganciclovir, or components of the product
- Inability to attend follow-up hearing and clinical assessments
- Infants with Auditory neuropathy/dyssynchrony.
- Children with another known etiology for SNHL (e.g. connexin 26, syndrome or metabolic disorder associated with SNHL, inner ear malformation and widened vestibular aqueducts, meningitis). Exclusion of each of these conditions is not required for trial enrollment.

## 4.4 Randomization and Blinding

(ICH E3; 9.4.3, 9.4.6. ICH E9; 2.3.1, 2.3.2)

The randomization schedule will be created by the UAB Data Coordinating Center (DCC).

Randomization will be implemented by the web-based randomization system developed and maintained at the UAB Data Coordinating Center at the University of Alabama at Birmingham. The generation and maintenance of study randomization codes will be the responsibility of the UAB Data Coordinating Center. The codes will be kept in a secure location in the Data Coordinating Center.

A site will enter the data via electronic data entry system (eDES). Once an eligible participant is enrolled, the subject's Guthrie card will be retrieved and tested for CMV DNA by PCR, unless there is a virologically confirmed diagnosis of congential CMV infection made within the first 30 days of life. Once a diagnosis of congenital infection is confirmed, the site will complete the Randomization form via eDES and will lock the form to successfully randomize a subject. Once the subject is randomized, an email alert will be sent to the site PI, site staff, and responsible parties containing information, randomization ID, center information and PK schematic for the subject. No information about the treatment assignment will be provided in this email alert. Site pharmacist will receive a separate email that contains the treatment assignment. Study monitors will be responsible for checking if the drug accountability documents shows the correct treatment based on the randomization email for each subject.

#### Blinding

Study subjects, investigators, and staff interacting with the study subjects will be masked to treatment. At the time of randomization, the site study pharmacist (who will not be masked to treatment) will prepare oral valganciclovir or oral placebo for distribution to the study subject. To ensure masking of all other study staff and families, study drug will be dispensed in amber bottles, along with amber-colored syringes for drawing up all doses. Additionally, the central audiologist who

analyzes the audiology data will be masked to study assignment, as will all personnel at the UAB Central Unit (with the exception of the UAB Study Statistician).

Upon completion of the six month follow-up period for all study subjects, or if the study is stopped early for any reason, the study will be unmasked after all enrolled study participants have completed the Month 6 follow-up assessments and the database is frozen. In an emergency situation, in which knowledge of the treatment assignment will be used to reduce/remove an immediate hazard to a volunteer, the study PI and/or a local site PI will have the ability to access the treatment assignment. In this situation (emergency unblinding) the study/local PI must explain and justify the nature of the event that resulted in the decision to immediately unblind to the DMID Medical Monitor and the Protocol Chair as soon as possible. This justification will be documented as a protocol deviation, and the IRBs and regulatory agencies will be informed as is appropriate.

Unmasking/Unblinding may also occur when the safety of a study participant is in question. In non-emergency situations, a conference call will be held to determine whether or not unmasking of an individual study subject is necessary or appropriate. The conference call will include the Protocol Chair, Protocol Statistician, DMID Medical Monitor and Clinical Project Manager.

The DSMB access to unblinded data is to be determined and will be based on the charter. Two data reports will be generated for each DSMB meeting: Open reports (with blinded information), and Closed reports (with unblinded information). The Closed Report will be prepared by the Protocol Statistician. Open reports will be distributed to and reviewed by the Sponsor (NIAID/DMID) and the CASG CU, and will be distributed to Genetech, Inc. The Closed Reports will be distributed to the Sponsor's pharmacovigilance contractor, DMID Clinical Research Operations and Management System (CROMS), via e-mail as a password protected Adobe Acrobat document. The password will be sent in a separate email. DMID CROMS then will distribute the Closed Reports only to the DSMB and maintain the reports as access restricted files.

# 4.5 Study Variables

(ICH E3; 9.5.1. ICH E9; 2.2.2)

The following table summarizes the visit, visit windows and the information to be collected and evaluations to be done at each visit.

| | Enrollment | Day - (Window: Day -30 | Study Day | | | | | Study Month | |
|---|---|---|---|---|---|---|---|---|---|
| | (Window: Day –<br>90 to Day –1) | | 1<br>(day -3 | 14<br>(± 2 | 28<br>(± 2 | 42<br>(± 2 | 70<br>(± 4 | 4<br>(± 7 | 6<br>(± 7 |
| | | | to day | days) | days) | days) | days) | days) | days) |
| Following study enrollment, testing of<br>Guthrie card for CMV DNA by PCR (if<br>congenital CMV infection has not already<br>been documented during first month of<br>life) | Х | | | | | | | | |
| Confirmation of congenital CMV infection<br>by documentation during first month of life<br>or by PCR-positive Guthrie card | | Х | | | | | | | |
| Baseline demographics <sup>a</sup> | | X | | | | | | | |
| Hematology Safety Labs <sup>b</sup> | | | X | Х | Х | Х | Х | | |
| Chemistry Safety Labs <sup>c</sup> | | | Х | Х | Х | Х | Х | | |
| Weight and Length | | | Х | Х | Х | | | | |
| Adverse Event Assessment | | | Х | Х | Х | Х | Х | | |
| Concurrent Medications | | | Х | Х | Х | Х | Х | | |
| Updated results of any etiological investigations for SNHL | | | х | х | х | х | х | х | Х |
| Hearing Assessment | | X <sup>d</sup><br>Day -90 to Day -1 | | | | | | | X<br>14-30<br>days |
| Virology Specimens for CMV Viral Loade | | | Х | Х | Х | Х | Х | Х | Х |
| Ganciclovir Population Pharmacokineticsf | | | | Х | Х | Χ | | | |

# Statistical Analysis Plan

# STUDY TITLE: DMID 11-0069

| Valganciclovir vs. Placebo Administration <sup>9</sup> | • | | | | | | |
|---|---|---|---|---|---|---|---|
| Total volume of blood required | 2.0 mL | 2.25 | 2.25 | 2.25 | 2.0 | 0.5 | 0.5 |
| Total volume of blood required | 2.0 1112 | mL | mL | mL | mL | mL | mL |

#### Statistical Analysis Plan

#### STUDY TITLE: DMID 11-0069

- a) Baseline demographics and birth history consist of date of birth; gender; race; ethnicity; birth weight; length at birth, if available; head circumference at birth, if available; and gestational age at birth. Degree of CMV disease involvement consists of neuroimaging abnormalities if imaging was performed; petechiae at any time from birth through study randomization, if hotained; hepatomegaly at any time from birth through study randomization, if noted; splenomegaly at any time from birth through study randomization, if noted; CSF white blood cell count at any time from birth through study randomization, if obtained; CSF cMV PCR at any time from birth through study randomization, if performed; seizures at any time from birth through study randomization, if noted; elevated transaminases at any time from birth through study randomization, if obtained; elevated bilirubin at any time from birth through study randomization, if obtained; medical history and baseline conditions prior to study randomization, by body system, chorioretinitis, intrauterine growth restriction, urine CMV testing (e.g., viral culture, shell-vial culture, PCR) within 90 days prior to study enrollment, if obtained clinically
- b) WBC with differential, hemoglobin, Platelet enumeration (approximate total blood needed for these tests is 0.5 mL)
- c) ALT, total bilirubin, creatinine (approximate total blood needed for these tests is 1.0 mL)
- d) BSER and/or VRA (to assess neuro-otologic status) and OAEs will be obtained. If the BSER and/or VRA is abnormal, then bone conduction will be obtained to distinguish between sensorineural hearing loss, conductive loss, and mixed loss. If the OAEs are abnormal, then acoustic immittance measures (tympanometry and acoustic reflexes) will be obtained to better define the middle or inner ear abnormality (e.g., otitis media).
- e) Required amount of whole blood for quantitative CMV PCR is at least 0.5 mL. Urine collection by bagged or clean catch specimen for quantitative PCR. Saliva collection by polyester fiber-tipped swabs for quantitative PCR.
- f) Required amount of whole blood for plasma ganciclovir determination is at least 0.25 mL
- g) Valganciclovir or placebo administration begins on Day 1 of the study; study medication dose adjusted for weight change, if needed, at each study visit while on treatment

Hearing assessments at each time point and at each ear as well as the change in the best ear comparing Month 6 with baseline will be provided by a single Independent Audiologist (IA) who will interpret the audiology reports of all patients at all protocol–specified visits requiring hearing assessments. The IA will enter the data directly to the eDES.

Section 3.3 describes the derived variables and the techniques and rules used to obtain the transformed data that will be used in the analyses

# 5 Sample Size

(ICH E3; 9.7.2. ICH E9; 3.5)

The planned enrollment is 54 subjects. Dropouts and subjects with audiology assessments that are inadequate for study comparison will be replaced (up to 20%, or n=10).

A sample size of 54 (27 in each arm) has 90% power to detect a worsening of hearing from 40% to 8.0% in the treatment group based on analyzing two correlated binary outcomes with correlation coefficient of 0.55 at 2.5% level of significance (using PASS 2008 program).

#### 6 General Considerations

## 6.1 Timing of Analyses

The final analysis will be performed after all subjects have completed study participation, all subjects have been 100% monitored by an independent monitor, data quality check has been completed and the data base has been locked.

# 6.2 Analysis Populations

(ICH E3; 9.7.1, 11.4.2.5. ICH E9; 5.2)

All enrolled subjects will be included in the basic demographic and clinical summaries and analyses. Only subjects who took at least one dose of the blinded treatment and who have completed hearing assessment data at baseline and Month 6 will be included in the analyses of study outcomes that compare treatment groups based on the intention—to—treat (ITT). Safety analyses will be done on all participants enrolled in the study. Children who have completed the full six weeks SAP version 2.0 DMID 11–0069 Date of Version 14 August 2020 Page 19 of 48

STUDY TITLE: DMID 11-0069

of study medication and have hearing assessment data at baseline and Month 6 will be included in a per-protocol (PP) analysis of efficacy, which will be performed as a sensitivity analysis.

## 6.3 Covariates and Subgroups

(ICH E3; 9.7.1, 11.4.2.1. ICH E9; 5.7)

The primary outcome will be analyzed using logistic regression based on generalized estimating equations (GEE) in order to accommodate the correlation between the left and right ears of a subject in the modeling. In addition, if there are enough data available we will adjust the analyses by whether or not a subject at birth is asymptomatic or symptomatic from their congenital CMV infection. Additional analyses will be performed to adjust for age and site plus any imbalances in the demographic and clinical characteristics to determine if adding them to the model will impact the results.

# 6.4 Missing Data

(ICH E3; 9.7.1, 11.4.2.2. ICH E9;5.3. EMA Guideline on Missing Data in Confirmatory Clinical Trials)

Primary analyses will be done on the first 54 subjects recruited. If there were subjects enrolled as replacement for dropouts or missing outcome, these added subjects will be included in the secondary analyses.

For those with missing outcome due to missing baseline and/or Month 6 audiology (including dropouts), we will exclude them from the primary analysis. However, we will perform sensitivity analysis by replacing all missing data with "worsening" outcome.

# 6.5 Interim Analyses and Data Monitoring

(ICH E3; 9.7.1, 11.4.2.3. ICH E9; 4.1, FDA Feb 2010 "Guidance for Industry Adaptive Design Clinical Trials for Drugs and Biologics")

No interim analysis for futility or efficacy is proposed because this is a small sample study and the penalty for an early look at the outcome data would compromise the study. However, a safety review will be done periodically.

#### 6.5.1 Safety Review

Safety reports will be generated and sent to DMID to be disseminated to the DSMB. This report includes hematology and safety laboratory values and adverse events (serious and non-serious). In addition, Section 9.7 provides a table of halting rules based on the number of subjects experiencing Grade 3 or 4 neutropenia for consideration by the DSMB.

## 6.5.2 Stopping Rules

In prior CASG studies of ganciclovir and valganciclovir that have enrolled 233 subjects, the only laboratory toxicity statistically associated with antiviral treatment has been neutropenia. Halting rules for this study therefore have been constructed to interrupt study enrollment if an excessive number of subjects are experiencing neutropenia. In the CASG 102 study, 63% of subjects receiving parenteral ganciclovir developed Grade 3 or Grade 4 neutropenia. In the CASG 109 study, 38% of subjects receiving oral valganciclovir developed Grade 3 or Grade 4 neutropenia.<sup>2</sup> Whether this lower rate of neutropenia relates to the mode of drug delivery is not known at this time. Assuming that 75% of subjects receiving ganciclovir developed Grade 3 or 4 neutropenia and given that randomization is expected to be balanced between those in study drug and those in placebo, the stopping rule will be based on assuming that the overall event rate for all study participants (i.e., placebo and active subjects combined) is 37.5%. Therefore, study enrollment will be stopped and an ad hoc review will be performed if a significantly higher proportion (37.5%) of subjects in this study experience Grade 3 or Grade 4 neutropenia, as detailed in the following table:

The stopping rules are based on the tail probabilities of the cumulative binomial. If the number of subjects "X" who experience Grade 3 or 4 neutropenia is greater than or equal to "m" out of "n" subjects, enrollment into the protocol will be held as described above while the DSMB decides whether study closure should occur. The stopping rules are based on the upper tail probabilities of the cumulative binomial with probability of an event set at 0.375. The cut-off numbers were determined by obtaining the largest value such that the tail probability is less than but closest to

0.05. More specifically, the following values of (m/n) apply for this Phase II protocol:

| | Stop/Investigate<br>when number with | Probability of observing X or more events | | Stop/Investigate when | Probability of observing X or more events |
|---|---|---|---|---|---|
| Number<br>enrolled (Y) | events equals this<br>number (X) | assuming<br>p=0.375 | Number<br>enrolled (Y) | number with events equals this number (X) | assuming p=0.375 |
| 4 | 4 | 0.020 | 30 | 17 | 0.025 |
| 5 | 5 | 0.007 | 31 | 17 | 0.037 |
| 6 | 5 | 0.031 | 32 | 18 | 0.024 |
| 7 | 6 | 0.013 | 33 | 18 | 0.034 |
| 8 | 6 | 0.036 | 34 | 18 | 0.048 |
| 9 | 7 | 0.017 | 35 | 19 | 0.032 |
| 10 | 7 | 0.038 | 36 | 19 | 0.044 |
| 11 | 8 | 0.019 | 37 | 20 | 0.030 |
| 12 | 8 | 0.039 | 38 | 20 | 0.041 |
| 13 | 9 | 0.021 | 39 | 21 | 0.028 |
| 14 | 9 | 0.039 | 40 | 21 | 0.038 |
| 15 | 10 | 0.021 | 41 | 22 | 0.026 |
| 16 | 10 | 0.037 | 42 | 22 | 0.035 |
| 17 | 11 | 0.021 | 43 | 22 | 0.047 |
| 18 | 11 | 0.036 | 44 | 23 | 0.032 |
| 19 | 12 | 0.021 | 45 | 23 | 0.043 |
| 20 | 12 | 0.034 | 46 | 24 | 0.030 |
| 21 | 13 | 0.020 | 47 | 24 | 0.040 |
| 22 | 13 | 0.033 | 48 | 25 | 0.028 |
| 23 | 13 | 0.050 | 49 | 25 | 0.037 |
| 24 | 14 | 0.031 | 50 | 25 | 0.048 |
| 25 | 14 | 0.046 | 51 | 26 | 0.034 |
| 26 | 15 | 0.029 | 52 | 26 | 0.044 |
| 27 | 15 | 0.043 | 53 | 27 | 0.032 |
| 28 | 16 | 0.027 | 54 | 27 | 0.041 |
| 29 | 16 | 0.040 | | | |

# 6.5.3 Adjustment of Confidence Intervals and p-values

STUDY TITLE: DMID 11-0069

There will be no planned adjustments on the confidence intervals since there is no proposed interim analysis.

#### 6.5.4 Practical Measures to Minimize Bias

Not applicable as there is no interim analysis for this study.

#### 6.5.5 Documentation of Interim Analyses

Not applicable as there is no interim analysis for this study

#### 6.6 Multi-center Studies

(ICH E3;9.7.1, 11.4.2.4. ICH E9; 3.2)

This study is a multi-center study. The primary outcome of hearing was analyzed by a single independent audiologist. Data will be analyzed by combining data from all study centers.

# 6.7 Multiple Testing

(ICH E3; 9.7.1, 11.4.2.5. ICH E9; 2.2.5)

Based on the hearing assessment of each ear at Month 6 and at Baseline, change in each ear will be categorized into binary outcome: improved + no change versus other (i.e. worsened). For example, normal in the left ear at baseline and moderate in the same ear at Month 6 will be considered as worsened. P-values < 0.05 will be considered significant for the primary outcomes. There are no planned adjustments for multiple testing for secondary outcomes.

# 7 Summary of Study Data

All continuous variables will be summarized using the following descriptive statistics: n (non-missing sample size), mean, standard error, median, maximum and minimum. The frequency and percentages (based on the non-missing sample size) of observed levels will be reported for all categorical measures. In general, all data will be listed, sorted by site, treatment and subject, and when appropriate by visit number within subject. All summary tables will be structured with a column for 1. Randomized/not randomized/total and 2. Active, placebo and total, and will be annotated with the total population size relevant to that table/treatment, including any missing observations.

# 7.1 Subject Disposition

The following flowchart will be used to summarize the subject disposition in the study and treatment. Numbers will be obtained based on the following CRFs: Inclusion/Exclusion, Randomization, Study Treatment Termination or Completion, and Study Termination or Completion.



Figure 2b: Treatment Disposition of Subjects



#### 7.2 Protocol Deviations

Protocol deviations will be summarized by site and type of deviation; deviations that resulted in adverse and serious adverse events; and protocol deviations that resulted in termination. The summary statistics will be produced in accordance with Section 7.

A raw listing of all protocol deviations will be provided by site by subject ID, deviation date, resulting in AE, SAE, and termination; deviation description; reason for the deviation; deviation category; effect on product stability; and deviation resolution.

As per protocol, if a study subject proceeds to cochlear implantation during the course of the study, he/she will not require additional study-related hearing assessments following the implantation procedure. Hence, hearing outcomes from these subjects past implantation will not be included in the analyses.

Finally, any subjects enrolled but not eligible will also be excluded from the analyses.

# 7.3 Demographic and Baseline Variables

- Age at enrollment (actual and categorized as 1-11 months, 12-23 months, 24-35 months, 36 or more months)
- Gender
- Ethnicity
- Gestational Age (actual and categorized as pre-term, i.e., 31-<=37 weeks, and term)
- Race
- Sex
- Birth Weight
- Length at birth
- Head circumference at birth

The summary statistics will be produced in accordance with section 7.

# 7.4 Degree of CMV Disease Involvement at Birth

The degree of CMV disease involvement at birth will be recorded, if known.

- Neuroimaging abnormalities
- Petechiae

- Thrombocytopenia
- Hepatomegaly
- Splenomegaly
- CSF white blood cell count
- CSF protein concentration
- CSF CMV PCR
- Seizures
- Elevated transaminases
- Elevated bilirubin

## 7.5 Concurrent Illnesses and Medical Conditions at Baseline

- Symptoms of CMV
- Medical and Surgical Abnormalities (Neurologic, Cardiovascular, Pulmonary, Gastrointestinal, HEENT, Musculoskeletal, Hepatobiliary/pancreatic, Hematologic/lymphatic, Genitourinary, Endocrine/metabolic, Dermatological, Immune system, Body as a whole, Metabolism and nutrition disorders)

STUDY TITLE: DMID 11-0069

• CMV disease involvement

The summary statistics will be produced in accordance with section 7.

#### 7.6 Prior and Concurrent Medications

Questions regarding medications will be asked at each visit. List of medications taken at baseline and at each visit, date medication started and stopped, or if medication being taken is ongoing will be noted. A listing by subject ID, visit, drug, start date, stop date, if ongoing or not, and reason for taking the medication will be provided. Summary of medications that were considered as prohibited medications while in the study will be presented as a separate listing.

## 7.7 Treatment Compliance

Ganciclovir plasma concentrations will be obtained with each blood draw obtained while the subject is receiving valganciclovir (Study Day 14, Study Day 28, and Study Day 42). For each subject, one of these three draws will occur 0 to 4 hours after a valganciclovir dose, one will occur 4 to 8 hours after a valganciclovir dose, and one will occur 8 to 12 hours after a valganciclovir dose. The summary statistics will be produced in accordance with section 7.

An integrated pharmacokinetic-adherence measure (IPAM) will be applied to determine the degree of regimen adherence. Briefly, this unique approach will compare predicted drug concentrations (Cpred) with measured concentrations (Cobs) to determine the magnitude of variability at each time point. A pharmacokinetic model will be developed for GCV. This model was used to simulate, or predict, the concentration that was measured in the subject at each clinic visit where a sample was obtained. If the log of Cpred/Cobs ratios clustered around zero, then the subject will be relatively adherent. If the log ratios will be consistent but deviated from zero, the subject was regularly non-adherent. Lastly, if the log ratios deviated widely from zero, the subject will exhibit a large degree of nonadherence. When the plausible sources of variability in plasma concentrations (i.e. pharmacokinetic, analytical, draw timing, and dosing history) will be considered, an acceptable range of difference between Cpred and Cobs will be approximately 40%. The number of Cobs that fell within this  $\pm 40\%$  range will be simply divided by the total number of observations to derive the IPAM score (e.g., 4 out of 8 samples within the range of variability equals 0.50 (50%) adherence). This will be done for 40%, 50%, and 60% variability. The IPAM score is therefore a continuous scale from 0.0 to 1.0. The average IPAM score for all subjects will be used to determine adherence rates relative to clinical outcomes and toxicities seen throughout the study period.

The summary statistics will be produced in accordance with section 7.

# 8 Efficacy Analyses

All efficacy variables will be listed by subject. Data will be summarized by treatment group. Continuous efficacy variables will be summarized by n, mean, standard error, minimum and maximum, and categorical efficacy variables will be summarized by number and percent.

# 8.1 Primary Efficacy Analysis

The primary endpoint is the change in total ear hearing assessments between baseline and 6 months, and will be assessed using the intent-to-treat population. At baseline and at 6 months, hearing thresholds (in decibels) will be determined using age-appropriate and developmentally-appropriate audiologic assessments. The decibel hearing thresholds in each ear classified whether the ear has normal hearing, mild hearing loss, moderate hearing loss, or severe hearing loss. Based on the hearing assessment of each ear at Month 6 and at Baseline, change in each ear

will be categorized into binary outcomes: improved or no change versus other. For example, normal in the left ear at baseline and moderate in the same ear at Month 6 will be considered as worsened. This binary outcome will be analyzed using logistic regression based on generalized estimating equations (GEE) in order to accommodate the correlation between the left and right ears of a subject in the modeling. In addition, if there are enough data available we will adjust the analyses by whether or not a subject at birth is asymptomatic or symptomatic from their congenital CMV infection. Additional analyses will be performed to adjust for age and site plus any imbalances in the demographic and clinical characteristics to determine if adding them to the model will impact the results. P-values < 0.05 will be considered significant for the primary outcomes.

A single, independent study audiologist who is masked (blinded) to treatment assignment will assess the audiology test battery for each subject and assign the classifications of normal hearing, mild hearing loss, moderate hearing loss, or severe hearing loss based upon their hearing thresholds (in decibels). The classifications will be assigned by ear (one for the left ear and one for the right ear), giving "total ear" classifications. , At the analyses stage, the "best ear" classification for the subject at that study visit will be determined; for example, if a subject had mild hearing loss in their left ear and severe hearing loss in their right ear, then the "best ear" classification will be mild hearing loss.

Primary analyses will be done on the first 54 subjects recruited. If there were subjects enrolled as replacement for dropouts or missing outcome, these added subjects will be included in the secondary analyses.

For those with missing outcome due to missing baseline and/or Month 6 audiology (including dropouts), we will exclude them from the primary analysis. However, we will perform sensitivity analysis by replacing all missing data with "worsening" outcome.

For those study subjects proceeding to cochlear implantation during the course of the study, he/she will not require additional study-related hearing assessments following the implantation procedure. Efficacy analyses will utilize "severe" as final hearing assessment at Month 6 for those who underwent cochlear implantation.

The summary statistics will be produced in accordance with section 7.

# 8.2 Secondary Efficacy Analyses

Logistic analyses will be utilized to determine if there is treatment effect based on the best ear outcome. As in the total ear analysis, change in the best ear will be categorized into binary outcomes – namely: improved + no change versus worse; improved + no change (normal to normal) versus worse + no change (abnormal to

abnormal); and improved versus other between baseline and Study Month 6. In addition to the primary outcome, we will analyze the binary outcome for change in the total ears categorized as: improved+ no change (normal to normal) versus worse and improved vs other.

For other secondary and tertiary outcomes, Fisher's exact test will be used to compare binary outcomes (such as detection of viruria or subject with at least one AE or SAE), and Wilcoxon Rank test will be used to compare continuous outcomes (such as quantitative log reduction) between the two treatment groups 6 weeks and 6 months after initial treatment.

Logistic model utilizing generalized estimating equations will also be used to determine the association between change in hearing and change in viral load. Change in viral load over time will be measured by the area under the curve computed using the trapezoidal rule. Spearman rank correlation will be utilized to examine the association between viral load and PK parameters. Poisson regression model will be used to compare the number of AEs/SAEs experienced by subjects between the two groups.

As in the primary outcomes, missing change in hearing outcomes will be replaced by worsened outcomes as sensitivity analyses for all secondary hearing outcomes.

The summary statistics will be produced in accordance with section 7.

# 9 Safety Analyses

Analyses of safety data will be based on data from all subjects receiving at least one dose of study drug. As per protocol, safety data will be collected only through Study Day 70, i.e., four weeks after the last study dose.

Incidence of serious and non-serious adverse events will be summarized by body system and system organ class using Medical Dictionary of Regulatory Activities (MedDRA) codes, the United States Division of AIDS (DAIDS) toxicity grade, and relation to drug. Frequencies (numbers and percentages) of subjects with one or more adverse events will be summarized by treatment group. Incidence of neutropenia and the incidence of adverse events leading to discontinuation of therapy will be assessed. Fisher's exact test will be used to compare proportions and Wilcoxon rank sum test will be used to compare continuous safety parameters

between two groups. Poisson regression model will be used to compare the number of AEs experienced by subjects between two groups.

Raw listings of all AEs and SAEs will be provided sorted by treatment group, subject ID and onset date.

When calculating the incidence of AEs by toxicity grade for a given body system, the most severe AE will be counted for subjects with multiple AEs.

# 9.1 Extent of Exposure

An integrated pharmacokinetic-adherence measure (IPAM) will be applied to determine the degree of regimen adherence (see Section 7.6 Treatment Compliance) for more details. In addition, ganciclovir concentration from PK analysis will be reported.

#### 9.2 Adverse Events

Analyses of AEs will be based on data from all subjects receiving at least one dose of study drug. As per protocol, safety data will be collected only through Study Day 70, i.e., four weeks after the last study dose.

AEs will be reported by treatment based on the relation to study drug, toxicity grade, and body system. When calculating the incidence of adverse events, or any sub-classification thereof by treatment, time period, severity, etc., each subject will only be counted once and any repetitions of adverse events will be ignored; the denominator will be the total number in each treatment group or overall sample size as appropriate.

# 9.3 Deaths, Serious Adverse Events and other Significant Adverse Events

Analyses of SAEs will be based on data from all subjects receiving at least one dose of study drug. As per protocol, safety data will be collected from Study Day 1 through four weeks following the last dose of study drug.

#### 9.4 Pregnancies

Not applicable to this study.

# 9.5 Clinical Laboratory Evaluations

STUDY TITLE: DMID 11-0069

Chemistry and hematology laboratory evaluations will be reported. The summary statistics will be produced in accordance with section 7. Flags are defined as values outside of the site- and age-specific normal ranges. The reported upper and lower limits by the site will be used to determine if the reported laboratory value was outside of the reported limits which will translate to a flag for the particular laboratory values. The number and percent (relative to the total laboratory done for that parameter) of flags will be reported in summary tables for each of the laboratory parameters. Means and standard errors of critical safety laboratory parameters (ANC, hemoglobin, WBC, platelet, ALT, bilirubin, and creatinine) over time will be displayed in a figure. Mixed model with random intercept and time, therapy and time by therapy interaction term will be will be used to compare the safety parameter at each time point between the treatment groups.

# 9.6 Other Safety Measures

Growth parameters (weight and length) will be captured serially. Fisher's exact test will be used to compare proportions and Wilcoxon rank sum test will be used to compare continuous safety parameters between two groups at each visit. Growth parameters will be presented graphically to monitor trends and compared at each time point for possible differences. The summary statistics will be produced in accordance with section 7.

#### 10 Pharmacokinetics

If the final number of usable PK specimens warrants, a population PK model may be applied to the dataset. The population PK modeling will be conducted using ADAPT 5 version 049.exe (Biomedical Simulations Resource, Los Angeles, CA), installed on a Dell Latitude E6410 laptop running Windows 7.0, 64 bit operating system( Intel Visual Fortran Compiler Professional Edition 11.1.070 Update 8 for Windows and Intel Math Kernel Library 10.2 Update 7 for Windows). For the analysis, all time values will be truncated. Instead of entering 6 weeks of dosing information, the timeline will be reduced to generally within 3–5 days depending upon the number of available concentration–time points for each subject. Thus, all samples will be still at steady–state. Population PK analysis will be conducted via a nonlinear mixed–effect model approach using ADAPT 5. The Maximum Likelihood Estimation Maximization (MLEM) algorithm will be used for all analyses. The PK base model will be identified previously as a one–compartment model with first–order input and

STUDY TITLE: DMID 11-0069

elimination. All inter-individual error terms in the PK parameters will be assumed to have a log-normal distribution. One error variance model will be used:

$$\operatorname{var}\left\{e\left(t\right)\right\} = \left(\sigma_{inter} + \sigma_{slope}y\left(t\right)\right)^{2}$$

where the proportional error model is SDslope and the additive error model is (SDinter). This is the most common error variance model used in ADAPT.

Model selection will be driven by the data and will be based on various goodness of fit indicators, including comparisons based on the Akaike information criteria (AIC), visual inspection of diagnostic scatter plots and evaluation of relative standard errors for the parameter and population estimates. Individual covariate assessments and a stepwise forward inclusion procedure ( $\alpha = 0.01$ ; i.e. the decrease of  $-2 \log 1$ likelihood [-2LL] values larger than 6.63) will be performed in ADAPT to build the full model. During the model building process, if the effects of two covariates will be highly correlated (such as weight and age), it may not have been possible to include both covariates into the model. In this case, in general, the variable with the highest significance (i.e., largest decrease in -2LL values from the base model) will be preferred, but when the decrease in -2LL will be very similar, clinical judgment may have been used to select which of the correlated covariates to include in the model. Covariate effects will be assumed to be linear based on visual inspection between each covariate and the PK parameter of interest (either CL/F and/or V/F). This analysis approach is similar to the analyses of the previous CASG 102 and 109 studies.

The summary statistics will be produced in accordance with section 7.

# 11 Virology

CMV whole blood viral load will be assessed by PCR at each study visit to assess for changes in viral load over time in study subjects with increasing whole blood viral loads during the course of treatment. Association of changes in whole blood viral load with changes in hearing between baseline and Study Month 6 in total ear and best ear will be evaluated as secondary endpoints. Change in the viral load over time will be measured by computing the average area under the curve (using trapezoidal rule) of all available viral load data for each subject, thus providing one

single value per participant. The area under the curve will be computed based on log base 10 viral load.

Hearing outcomes for this correlation analyses will be based on change in total ear from baseline to Study Month 6. The primary outcome will be defined with regard to change in the total ear: improved or no change versus other (i.e., worsened). Logistic regression based on generalized estimating equations will be utilized to assess if change in the viral load will be associated with the change in the total ear hearing outcomes in order to account for the correlation between outcomes attributed to the left and right ear for the same subject.

All the comments from section 7 onwards may be relevant.

# 12 Figures

Figures will be used to represent the following:

- enrollment status
- rate of enrollment
- trends of growth parameters (weight and length) over time
- critical safety laboratory parameters (ANC, hemoglobin, WBC, platelet, ALT, bilirubin, and creatinine) over time
- display the study visit flow
- study disposition
- extent of exposure to treatment; ganciclovir concentration over time
- dosage over time
- log base 10 viral load over time
- audiology assessment available at baseline and Month 6.

# 13 Reporting Conventions

P-values will be reported to 4 decimal places. The mean, standard errors, and any other statistics other than quantiles, will be reported to one decimal

place. Quantiles, such as median, or minimum and maximum will use the same number of decimal places as the original data. Estimated parameters, not on the same scale as raw observations (e.g. regression coefficients) will be reported to 3 significant figures.

#### 14 Technical Details

A second review statistician will independently reproduce the primary analyses and summary statistics tables listed below:

Table 9b: Frequency of Serious Adverse Events by Body System, Grade and Therapy Group

Table 10a: Frequency of Adverse Events by Therapy, Body System, and Grade\*

Table 10b: AE Grade by Therapy Group

Table 21a: Quality of Hearing Assessment Left and Right (Total Ear)

Table 21b: Hearing Assessment Left and Right (Total Ear)

Table 21c: Change in Total Ear Hearing at Month 6 Relative to Baseline

Table 21d: Results of Modeling Treatment Effect on Total Ear For Each Outcome

Table 21e: Subgroup Analysis (Total Ears)

Table 22a: Quality of Hearing Assessment Best Ear

Table 22b: Hearing Assessment Best Ear

Table 22c: Change in Best Ear Hearing at Month 6 Relative to Baseline

Table 22d: Results of Analyses of Treatment Effect on Best Ear For Each Outcome

Table 22e: Subgroup Analysis (Best Ears)

Table 23: CMV Detection Over time

Table 24: Log10 Viral Load Summary Statistics Over Time

Table 24a: Summary of Modeling Results (Blood)

Table 24b: Summary of Modeling Results (Saliva)

Table 24c: Summary of Modeling Results (Urine)

Table 25: Spearman Rank Correlation between GCV concentration and log10 VL

Table 26a: Summary Statistics: Baseline Log10 VL by Change in Total Ear Hearing

Table 26b: Association between Baseline Log10 VL and Change (Binary) in Total Ear Hearing

Table 27a: Summary Statistics: Baseline Log10 VL by Change in Best Ear Hearing

Table 27b: Association between Baseline Log10 VL and Change (Binary) in Best Ear Hearing
Table 28a: Summary Statistics: Average AUC Log10 VL and Change in Total Ear Hearing

Table 28b: Association between Average AUC Log10 VL and Change (Binary) in Total Ear Hearing

Table 29a: Summary Statistics: Average AUC Log10 VL and Change in Best Ear Hearing

Table 29b: Association between Average AUC Log10 VL and Change (Binary) in Best Ear Hearing

Table 30a: Summary Statistics: Change in Log10 VL and Change in Total Ear Hearing Table 30b: Association between Change in Log10 VL and Change (Binary) in Total Ear Hearing

Table 31a: Summary Statistics: Change in Log10 VL and Change in Best Ear Hearing Table 31b: Association between Change in Log10 VL and Change (Binary) in Best Ear Hearing

### 15 Summary of Changes to the Protocol

The first version of the protocol under which subjects may be enrolled was Version 3.0.

The protocol was revised to Version 4.0, dated April 28, 2016, which was distributed to the study sites on May 5, 2016 for submission to their IRBs. Under this protocol version, study inclusion criteria and study windows have been liberalized based on the specific screen failure data under earlier protocol versions. Specifically, the inclusion criterion, "CMV shedding in urine by PCR or culture (including shell vial) within 12 weeks prior to study enrollment" was removed; the window for the Baseline study visit was changed from "Day –3 to Day 1" to "Day –30 to Day 1"; the window for the baseline hearing assessment was changed from "Study Day –14 to Study Day 7" to "Study Day –90 to Study Day –1"; and the window for the Month 6 hearing assessment was changed from "± 14 days" to "–14 days to +30 days".

#### 16 References

1 Kimberlin DW, Lin CY, Sanchez PJ, et al. Effect of ganciclovir therapy on hearing in symptomatic congenital cytomegalovirus disease involving the central nervous system: a randomized, controlled trial. *J Pediatr*. 2003;143:16–25.

2 Kimberlin DW, Acosta EP, Sanchez PJ, et al. Pharmacokinetic and pharmacodynamic assessment of oral valganciclovir in the treatment of symptomatic congenital cytomegalovirus disease. *J Infect Dis.* 2008;197:836-45.

# 17 ting of Tables and Listings Figures

### LIST OF TABLES

| Table Title | Number | Population | Endpoint | Time Points or how to conglomerate | Covariates or Subgroups | Summary<br>Statistics | Formal Analysis |
|---|---|---|---|---|---|---|---|
| Table 1a: Investigators / Centers | 1a | NA | NA | NA | NA | Listing | NA |
| Table 1b: Randomization to<br>Blinded Therapy Groups | 1b | Randomized | NA | NA | Therapy Group | n, % | NA |
| Table 2a: Distribution of Subjects<br>by Study Site and Therapy<br>Group, and Overall | 2a | NA | NA | NA | NA | Listing | NA |
| Table 2b: Reasons for withdrawal before randomization | 2b | NA | NA | NA | NA | Listing | NA |
| Table 2c: Site Performance in Enrollment | 2c | NA | NA | NA | NA | Listing | NA |
| Table 3: Subjects Withdrawn after Randomization from Study | 3 | NA | NA | Randomization-<br>Month 6 | NA | Listing | NA |
| Table 4a: Subject-specific Protocol Deviations by Category | 4a | Full Analysis | Deviations | Baseline-Month6 | NA | Listing | NA |
| Table 4b: Subject-specific Protocol Deviations by Reason | 4b | Full Analysis | Deviations | Baseline-Month6 | NA | Listing | NA |
| Table 4c: Listing of Action/Steps:<br>Subject-specific PDs | 4c | Full Analysis | NA | Baseline-Month6 | NA | Listing | NA |
| Table 4d: Subject-Specific Protocol Deviations resulting in AEs, SAEs, termination or drug interruption in study drug | 4d | Full Analysis | Deviations | Baseline-Month6 | NA | Listing | NA |
| Table 5a: Site-specific Protocol<br>Deviations by Category and<br>Reasons | 5a | Full Analysis | Deviations | Baseline-Month6 | NA | Listing | NA |
| Table 5b: Listing of Action/Steps: site-specific PDs | 5b | Full Analysis | NA | Baseline-Month6 | NA | Listing | NA |
| Table 6a: Frequency Counts of Baseline Demographics | 6a | Full Analysis | Demographics | Baseline | Therapy Group | n, % | Fisher's exact |

| Table 6b: Summary Statistics of<br>Baseline Age, Gestational Age<br>and Birth Weight | 6b | Full Analysis | Age, Gestational<br>Age and Birth<br>Weight | Baseline | Therapy Group | N, N Missing,<br>Mean, SE,<br>Median, Min,<br>Max | T-test or Wilcoxon |
|---|---|---|---|---|---|---|---|
| Table 7a: Summary of frequency count of CMV disease involvement | 7a | Full Analysis | CMV disease involvement | Baseline | Therapy Group | n, % | Fisher's exact |
| Table 7b: Summary CMV disease involvement: Lumbar Puncture | 7b | Full Analysis<br>(where<br>available) | CMV disease involvement | Baseline | Therapy Group | n, % | Fisher's exact |
| Table 7c: Summary of CMV disease involvement: Neuroimaging Results | 7c | Full Analysis<br>(where<br>available) | CMV disease involvement | Baseline | Therapy Group | n, % | Fisher's exact |
| Table 7d: Summary of Baseline<br>Abnormal Findings | 7d | Full Analysis<br>(where<br>available) | Abnormality | Baseline | Therapy Group | n, % | Fisher's exact |
| Table 8a: Summary of Adverse<br>Events | 8a | At least one dose of study drug | Adverse Events | Randomization-<br>Day 70 | Therapy Group | n, % | NA |
| Table 9a: Listing of Each<br>Subject's Serious Adverse Event | 9a | At least one dose of study drug | Serious Adverse<br>Events | Randomization-<br>Day 70 | Therapy Group | Listing | NA |
| Table 9b: Frequency of Serious<br>Adverse Events by Body System,<br>Grade and Therapy Group | 9b | At least one dose of study drug | Serious Adverse<br>Events | Randomization-<br>Day 70 | Therapy Group, Body<br>System, Grade | n, % | NA |
| Table 10a: Frequency of Adverse<br>Events by Therapy, Body System,<br>and Grade* | 10a | At least one dose of study drug | Serious Adverse<br>Events | Randomization-<br>Day 70 | Therapy Group, Body<br>System, Grade | n, % | NA |
| Table 10b: AE Grade by Therapy<br>Group | 10b | At least one<br>dose of study<br>drug | Adverse Events | Randomization-<br>Day 70 | Therapy Group, Grade | n, % | generalized linear<br>mixed model for<br>ordinal response with<br>random intercept. |
| Table 10c: Listing of Adverse<br>Events (Active Group) | 10c | At least one dose of study drug | Adverse Events | Randomization-<br>Day 70 | NA | Listing | NA |
| Table 10c: Listing of Adverse<br>Events (Placebo Group) | 10c | At least one dose of study drug | Adverse Events | Randomization-<br>Day 70 | NA | Listing | NA |

| Table 11a: Changes over Time in<br>Hematology Parameters | 11a | At least one<br>dose of study<br>drug | Hematology<br>Parameters | Baseline-Month 6 | Therapy Group, Visit | N, Mean, SD,<br>10th pctl,<br>90th pctl | General linear mixed model with random intercept was fitted for each parameter. Each model contains therapy, time and therapy by time interaction. |
|---|---|---|---|---|---|---|---|
| Table 11b: Changes over Time in<br>Chemistry Parameters | 11b | At least one<br>dose of study<br>drug | Chemistry<br>Parameters | Baseline-Month 6 | Therapy Group, Visit | N, Mean, SD,<br>10th pctl,<br>90th pctl | General linear mixed model with random intercept was fitted for each parameter. Each model contains therapy, time and therapy by time interaction. |
| Table 12: Maximum Degree of<br>Neutropenia (Lowest ANC)<br>During Day 1-42 Period | 12 | At least one dose of study drug | ANC | Randomization-<br>Day 42 | Therapy Group | n, % | NA |
| Table 13: Maximum Degree of<br>Anemia (Lowest HGB) for 11-<br>0069 Valganciclovir | 13 | At least one<br>dose of study<br>drug | HGB | Randomization-<br>Day 70 | NA | n, % | NA |
| Table 14: Maximum Degree of<br>Anemia (Lowest PLT) for 11-<br>0069 Valganciclovir | 14 | At least one dose of study drug | PLT | Randomization-<br>Day 70 | NA | n, % | NA |
| Table 15: Maximum Degree of<br>ALT (Highest ALT) for 11-0069<br>Valganciclovir | 15 | At least one dose of study drug | ALT | Randomization-<br>Day 70 | NA | n, % | NA |
| Table 16: Maximum Degree of<br>Creatinine (Highest creatinine)<br>for 11-0069 Valganciclovir | 16 | At least one<br>dose of study<br>drug | creatinine | Randomization-<br>Day 70 | NA | n, % | NA |
| Table 17: Summary of Concomitant Medications by Treatment Group (Blinded Treatment Phase) | 17 | At least one<br>dose of study<br>drug | Treatment<br>Group (Blinded<br>Treatment Phase | Baseline-Day 48 | Therapy Group, Visit | n, % | NA |
| Table 18a: Dose (mg/kg) of<br>Valganciclovir or Placebo | 18a | At least one<br>dose of study<br>drug | Dose | Day 1, 14 28 | Therapy Group, Visit | N, Mean, SD,<br>Median, Min,<br>Max | Fisher's exact and<br>Wilcoxon test |

| Table 18b: Weight (kg) at the Time of Dosing of Valganciclovir or Placebo | 18b | At least one<br>dose of study<br>drug | Dose | Day 1, 14 28 | Therapy Group, Visit | N, Mean, SD,<br>Median, Min,<br>Max | General linear mixed model with random intercept was fitted for each parameter. Each model contains therapy, time and therapy by time interaction. |
|---|---|---|---|---|---|---|---|
| Table 18c: Length (cm) at the<br>Time of Dosing of Valganciclovir<br>or Placebo | 18c | At least one<br>dose of study<br>drug | Weight | Day 1, 14 28 | Therapy Group, Visit | N, Mean, SD,<br>Median, Min,<br>Max | General linear mixed model with random intercept was fitted for each parameter. Each model contains therapy, time and therapy by time interaction. |
| Table 19a: Dosing Administration by Treatment Group and Visit | 19 | At least one dose of study drug | Length | Day 1, 14 28 | Therapy Group, Visit | n, % | Fisher's exact |
| Table 19b: Reasons for Adjusted or Held Dose and Significant Changes in Laboratory Parameters | 19a | At least one<br>dose of study<br>drug | Dose | Day 1, 14 28 | Therapy Group, Visit | n, % | Fisher's exact |
| Table 20: PK Specimen Results:<br>GCV concentration in the Active<br>Group | 19b | At least one<br>dose of study<br>drug | Dose | Day 1, 14 28 | NA | N, Mean, SD,<br>Median, Min,<br>Max | NA |
| Table 21a: Quality of Hearing<br>Assessment Left and Right (Total<br>Ear) | 20 | At least one<br>dose of study<br>drug | GCV<br>concentration | Day 14, 28, 42 | NA | n, % | NA |
| Table 21b: Hearing Assessment<br>Left and Right (Total Ear) | 21a | At least one dose of study drug | Quality of Total<br>Ear Assessment | Baseline and<br>Month 6 | Therapy Group, Visit | n, % | NA |
| Table 21c: Change in Total Ear<br>Hearing at Month 6 Relative to<br>Baseline | 21b | At least one<br>dose of study<br>drug | Hearing<br>Assessment<br>Total Ear | Baseline and<br>Month 6 | Therapy Group, Visit | n, % | NA |

| Table 21d: Results of Modeling<br>Treatment Effect on Total Ear<br>For Each Outcome | 21c | At least one<br>dose of study<br>drug | Change in Total<br>Ear Hearing<br>Assessment | Baseline and<br>Month 6 | Therapy Group | n, %, p-value | Generalized linear model for binary outcome using GEE was fitted for each parameter. Each model contains therapy, time and therapy by time interaction. |
|---|---|---|---|---|---|---|---|
| Table 21e: Subgroup Analysis<br>(Total Ears) | 21d | At least one dose of study drug | Change in Total<br>Ear Hearing<br>Assessment | Baseline and<br>Month 6 | Therapy Group | n, % | NA |
| Table 22a: Quality of Hearing<br>Assessment Best Ear | 21e | At least one dose of study drug | Change in Total<br>Ear Hearing<br>Assessment | Baseline and<br>Month 6 | Therapy Group | n, % | NA |
| Table 22b: Hearing Assessment<br>Best Ear | 22a | At least one dose of study drug | Quality of Best<br>Ear Assessment | Baseline and<br>Month 6 | Therapy Group | n, % | NA |
| Table 22c: Change in Best Ear<br>Hearing at Month 6 Relative to<br>Baseline | 22b | At least one dose of study drug | Hearing<br>Assessment Best<br>Ear | Baseline and<br>Month 6 | Therapy Group | n, % | NA |
| Table 22d: Results of Analyses of<br>Treatment Effect on Best Ear For<br>Each Outcome | 22c | At least one<br>dose of study<br>drug | Change in Best<br>Ear Hearing<br>Assessment | Baseline and<br>Month 6 | Therapy Group | n, %, p-value | Generalized linear model for binary outcome using GEE was fitted for each parameter. Each model contains therapy, time and therapy by time interaction. |
| Table 22e: Subgroup Analysis<br>(Best Ears) | 22d | At least one<br>dose of study<br>drug | Change in Best<br>Ear Hearing<br>Assessment | Baseline and<br>Month 6 | Therapy Group, Visit (age and symptomatic/asymptomatic at birth) | n, % | NA |
| Table 23: CMV Detection Over time | 22e | At least one dose of study drug | Change in Best<br>Ear Hearing<br>Assessment | Baseline and<br>Month 6 | Therapy Group, Visit | n, %, p-value | Fisher's exact |
| Table 24: Log10 Viral Load<br>Summary Statistics Over Time | 23 | At least one dose of study drug | CMV detection | Baseline-Month6 | Therapy Group, Visit | N, Mean, SD,<br>10th pctl,<br>90th pctl | NA |

| Table 24a: Summary of<br>Modeling Results (Blood) | 24 | At least one<br>dose of study<br>drug | Quantitative<br>Viral Load | Baseline-Month6 | Therapy Group, Visit | p-value | General linear mixed model with random intercept was fitted for each parameter. Each model contains therapy, time and therapy by time interaction. |
|---|---|---|---|---|---|---|---|
| Table 24b: Summary of<br>Modeling Results (Saliva) | 24a | At least one<br>dose of study<br>drug | Quantitative<br>Viral Load<br>(Blood) | Baseline-Month6 | Therapy Group, Visit | p-value | General linear mixed model with random intercept was fitted for each parameter. Each model contains therapy, time and therapy by time interaction. |
| Table 24c: Summary of Modeling<br>Results (Urine) | 24b | At least one<br>dose of study<br>drug | Quantitative<br>Viral Load<br>(Saliva) | Baseline-Month6 | Therapy Group, Visit | p-value | General linear mixed model with random intercept was fitted for each parameter. Each model contains therapy, time and therapy by time interaction. |
| Table 25: Spearman Rank Correlation between GCV concentration and log10 VL | 24c | At least one dose of study drug | Quantitative<br>Viral Load<br>(Urine) | Day 14, 28, 42 | NA | Correlation, p-<br>value | Spearman Rank<br>Correlation |
| Table 26a: Summary Statistics: Baseline Log10 VL by Change in Total Ear Hearing | 25 | At least one<br>dose of study<br>drug | concentration<br>and log10 VL | Baseline | Baseline Viral Load, Therapy<br>Group | N, Mean, SD,<br>10th pctl,<br>90th pctl | NA |
| Table 26b: Association between<br>Baseline Log10 VL and Change<br>(Binary) in Total Ear Hearing | 26a | At least one<br>dose of study<br>drug | VL by Change in<br>Total Ear Hearing | Baseline | Baseline Viral Load, Therapy<br>Group | N, Mean, SD,<br>10th pctl,<br>90th pctl with<br>p-values | Generalized linear model for binary outcome using generalized estimating equations with VL as main predictor for unadjusted model; adjusted model includes therapy group |

| Table 27a: Summary Statistics: Baseline Log10 VL by Change in Best Ear Hearing | 26b | At least one dose of study drug | VL and Change<br>(Binary | Baseline | Baseline Viral Load, Therapy<br>Group | N, Mean, SD,<br>10th pctl,<br>90th pctl | NA |
|---|---|---|---|---|---|---|---|
| Table 27b: Association between<br>Baseline Log10 VL and Change<br>(Binary) in Best Ear Hearing | 27a | At least one<br>dose of study<br>drug | VL by Change in<br>Best Ear Hearing | Baseline | Baseline Viral Load, Therapy<br>Group | N, Mean, SD,<br>10th pctl,<br>90th pctl with<br>p-values | Generalized linear<br>model for binary<br>outcome using<br>generalized estimating<br>equations with VL as<br>main predictor for<br>unadjusted model;<br>adjusted model<br>includes therapy group |
| Table 28a: Summary Statistics: Average AUC Log10 VL and Change in Total Ear Hearing | 27b | At least one<br>dose of study<br>drug | VL and Change<br>(Binary | Baseline-Month6 | AUC Viral Load, Therapy<br>Group | N, Mean, SD,<br>10th pctl,<br>90th pctl | NA |
| Table 28b: Association between<br>Average AUC Log10 VL and<br>Change (Binary) in Total Ear<br>Hearing | 28a | At least one<br>dose of study<br>drug | Log10 VL and<br>Change in Total<br>Ear Hearing | Baseline-Month6 | AUC Viral Load, Therapy<br>Group | N, Mean, SD,<br>10th pctl,<br>90th pctl with<br>p-values | Generalized linear<br>model for binary<br>outcome using<br>generalized estimating<br>equations with VL as<br>main predictor for<br>unadjusted model;<br>adjusted model<br>includes therapy group |
| Table 29a: Summary Statistics: Average AUC Log10 VL and Change in Best Ear Hearing | 28b | At least one dose of study drug | Log10 VL and<br>Change (Binary | Baseline-Month6 | AUC Viral Load, Therapy<br>Group | N, Mean, SD,<br>10th pctl,<br>90th pctl | NA |
| Table 29b: Association between<br>Average AUC Log10 VL and<br>Change (Binary) in Best Ear<br>Hearing | 29a | At least one<br>dose of study<br>drug | Log10 VL and<br>Change in Best<br>Ear Hearing | Baseline-Month6 | AUC Viral Load, Therapy<br>Group | N, Mean, SD,<br>10th pctl,<br>90th pctl with<br>p-values | Generalized linear model for binary outcome using generalized estimating equations with VL as main predictor for unadjusted model; adjusted model includes therapy group |
| Table 30a: Summary Statistics:<br>Change in Log10 VL and Change<br>in Total Ear Hearing | 29b | At least one<br>dose of study<br>drug | Log10 VL and<br>Change (Binary | Baseline-Month6 | Difference in Viral Load,<br>Therapy Group | N, Mean, SD,<br>10th pctl,<br>90th pctl | NA |

#### STUDY TITLE: DMID 11-0069

| Table 30b: Association between<br>Change in Log10 VL and Change<br>(Binary) in Total Ear Hearing | 30a | At least one<br>dose of study<br>drug | Log10 VL and<br>Change in Total<br>Ear Hearing | Baseline-Month6 | Difference in Viral Load,<br>Therapy Group | N, Mean, SD,<br>10th pctl,<br>90th pctl with<br>p-values | Generalized linear<br>model for binary<br>outcome using<br>generalized estimating<br>equations with VL as<br>main predictor for<br>unadjusted model;<br>adjusted model<br>includes therapy group |
|---|---|---|---|---|---|---|---|
| Table 31a: Summary Statistics:<br>Change in Log10 VL and Change<br>in Best Ear Hearing | 30b | At least one dose of study drug | Log10 VL and<br>Change (Binary | Baseline-Month6 | Difference in Viral Load,<br>Therapy Group | N, Mean, SD,<br>10th pctl,<br>90th pctl | NA |
| Table 31b: Association between<br>Change in Log10 VL and Change<br>(Binary) in Best Ear Hearing | 31a | At least one<br>dose of study<br>drug | Log10 VL and<br>Change in Best<br>Ear Hearing | Baseline-Month6 | Difference in Viral Load,<br>Therapy Group | N, Mean, SD,<br>10th pctl,<br>90th pctl with<br>p-values | Generalized linear model for binary outcome using generalized estimating equations with VL as main predictor for unadjusted model; adjusted model includes therapy group |

#### LIST OF FIGURES

Figure 1: Participant Flow Diagram

Figure 2: Rate of Enrollment

Figure 3a: Disposition of Subjects with Study Drug Information

Figure 3b: Disposition of Randomized Subjects with Study Drug Information

Figure 4: Changes in Hematology Parameters over Time for Enrolled Subjects

Figure 4a: Plot of WBC mean (±SE) over time

STUDY TITLE: DMID 11-0069

Figure 4b: Boxplots of WBC over time

Figure 4c: Plot of Hemoglobin mean (±SE) over time

Figure 4d: Boxplots of Hemoglobin over time

Figure 4e: Plot of ANC mean (±SE) over time

Figure 4f: Boxplots of ANC over time

Figure 4g: Plot of Platelet mean ( $\pm$ SE) over time

Figure 4h: Boxplots of Platelet over time

Figure 5: Changes in Chemistry Parameters over Time for Enrolled Subjects

Figure 5a: Plot of Serum Creatinine mean ( $\pm$ SE) over time

Figure 5b: Boxplots of Serum Creatinine over time

Figure 5c: Plot of Creatinine Clearance mean (±SE) over time

Figure 5d: Boxplots of Creatinine Clearance over time

Figure 5e: Plot of ALT mean (±SE) over time

Figure 5f: Boxplots of ALT over time

Figure 5g: Plot of Total Bilirubin mean (±SE) over time

Figure 5h: Boxplots of Total Bilirubin over time

Figure 6a: Dose (mg/kg) over Time

Figure 6b: Weight at Dosing

Figure 6c: Length (cm) at the Time of Dosing

Figure 7a: Change over Time in GCV concentration (linear scale)

Figure 7b: Change over Time in GCV concentration (Log scale)

Figure 8: Percent Detected Over Time

Figure 9a: Log 10 VL over time (Blood)

- Figure 9b: Log 10 VL over time (Saliva)
- Figure 9c.: Log 10 VL over time (Urine)
- Figure 10: Boxplots: Baseline Log10 VL and Change (Binary) in Total Ear Hearing
- Figure 11: Boxplots: Baseline Log10 VL and Change (Binary) in Best Ear Hearing
- Figure 12: Boxplots: Average AUC Log10 VL and Change (Binary) in Total Ear Hearing
- Figure 13: Boxplots: Average AUC Log10 VL and Change (Binary) in Best Ear Hearing
- Figure 14: Boxplots: Change in Log10 VL and Change (Binary) in Total Ear Hearing
- Figure 15: Boxplots: Change in Log10 VL and Change (Binary) in Best Ear Hearing

LISTINGS IN THE APPENDIX

- Appendix A: Hearing Assessment Listing
- Appendix B Specimen Shipment Tracking
- Appendix C: Concomitant Medications